CLINICAL TRIAL: NCT07325084
Title: Sustainable Football: Physical Profile, Training Load, Risk Factors and Injuries in Swedish Elite Football
Brief Title: Sustainable Elite Football
Status: Enrolling by invitation | Type: Observational
Sponsor: Linnaeus University (Other)
Responsible Party: Principal Investigator, Sofia Ryman Ryman Augustsson, Associate Professor, Linnaeus University
Other Study IDs: 2024-05136-01
Record Dates: First submitted 2024-11-04; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Overuse Injury; Traumatic Injury
Keywords: football; soccer; physical performance; injury risk factors
MeSH Terms: conditions — Cumulative Trauma Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Professional football players: 100 professional or semi-professional football players that plays in one of the two top division in Sweden.
- Academy football players: 300 academy football players between 15-19 years old.

SUMMARY:
The literature is scarce when it comes to more comprehensive research project that investigates the differences between youth and adult elite football players in physical parameters and the risk of injury. There is a lack of prospective long-term studies examining the importance of increased training load, physical fitness and performance, training status, position and maturity on its relationship to injury and success in elite football.

The aim of the project is to evaluate different aspects of physical performance, training load and their role as potential risk or protective factors for injury in elite Swedish football. Another aim is to follow youth players at the football academy to explore which physical factors are important for success in elite football and how a possible injury affects the player's continued elite efforts. Finally, the aim is to develop a test battery that can be used to screen for deficits in physical fitness, monitor football players at risk of injury and for return to sport after injury. The main research question intended to be investigated is: How do internal and external load, wellness, and physical performance factors (including Acute Chronic Workload Ratio) differ between academy-level and professional football players, and how do these factors relate to injury risk and success in elite football? A cohort design will be used with ~200 academy football players (~50% women) between 15-19 years old and 50 professional football players participating. The study starts with the assessment of different aspects of physical performance at baseline during the players first year at the academy and internal and external training load and injuries will be registered prospectively for 3 years. The players will be assessed at follow-ups, with the same tests, 3 times a year, to evaluate performance changes. Players who will be transferred to elite play will be evaluated 3 times a year for additional 5 years. Professional football players will also be evaluated with tests with following registration of training load and injuries.

DETAILED DESCRIPTION:
Purpose and aims

The aim of the project is to evaluate different aspects of physical fitness, muscle function, training load and their role as potential risk or protective factors for injury in elite Swedish football. Another aim is to follow youth players at the football academy (Swedish sports high schools for football) to explore which physical factors are important for success in elite football and how a possible injury affects the player's continued elite efforts. Finally, the aim is to develop a test battery that can be used to screen for deficits in physical fitness, monitor football players at risk of injury and for return to sport after injury. The following research questions are intended to be investigated:

1. What is the internal and external load and Acute Chronic Workload Ratio in football players at academy level compared to professional level?
2. What are the levels of wellness in football players at academy level compared to professional level?
3. Is impaired physical fitness and muscle function (physical performance) a risk factor for injury in football?
4. Which physical factors are important for success in elite football?
5. What impact has an injury on the youth player's continued elite efforts?
6. Can a test battery be used to screen for deficits in physical performance at the same time monitor football players at risk of injury?
7. Which physical factors are important for return to sport after injury in football?

Procedure and time frame The study is expected to begin with pilot testing in November 2024 and then set off in January 2025 with assessment of different aspects of physical performance at baseline during the players first year at the academy and internal and external training load and injuries will be registered prospectively for 3 years. The players will be assessed at follow-ups, with the same tests, 3 times a year, to evaluate performance changes. Players who will be transferred to elite play will be evaluated 3 times a year for additional 5 years. New academy players will take part in 2026 and 2027 following the same procedure. The professional football players will also be evaluated with tests with following registration of training load and injuries.

Measurements Injury registration Data on injury will be collected using a form7 distributed by the team's RPT. All players will report injuries occurring during sport activity diagnosed by a physical examination, MRI, or arthroscopy. Details on injury situation, and diagnosis will be reported by the team's RPT.

External and internal training load For the academy players, external training load will be collected weekly by reporting hours of match and training using a web-based form5 distributed through SurveyMonkey®. For the professional players external training load will be analyzed using data from the GPS system Polar Team Pro tracking devices. All players will also estimate session ratings of perceived exertion (sRPE) after each football session and Freshness score; muscle soreness, sleep quality and mental stress, before every session. Internal training load and Acute Chronic Workload Ratio (ACWR) will be calculated using sRPE multiplied by training minutes2.

Anthropometry Body height (cm) will be measured with a stadiometer, and body mass (kg) will be obtained from a bioelectrical impedance analysis (BIA) measurement (InBody 770, InBody Co, Ltd, Seoul, South Korea) together with total body lean body mass (LBM).

Physical Performance assessment The tests will be instructed and supervised by educated test leaders, and will take place at Slottslabbet, Radix, at Linnaeus University beginning with a warm-up protocol.

Jump performance Jump performance will be evaluated by the vertical jump test and performed as a counter-movement jump with the computerized system (MuscleLab, Ergotest Technology), as described8.

Squat strength Multiple joint maximal muscle strength of the lower extremity will be measured with the Isometric squat test, as described9. Peak isometric force (N) and avgRFD (N·s-1) are recorded and assessed using a force plate and analyzed with commercial software (MuscleLab, Ergotest Technology AS, Langesund, Norway).

Test of Nordic hamstring exercise (NHE) performance Both the fast stretch-shortening cycle and slow eccentric NHE will be measured using the protocol by Augustsson et al.9. During the NHEs, a linear encoder will be used to measure the position where the peak knee flexor force is recorded.

Isokinetic strength testing Strength testing of the quadriceps and hamstring muscles will be conducted unilaterally with players seated on an isokinetic dynamometer (Biodex System 4; Biodex Medical System), as described8 assessing both eccentric and concentric muscle actions. Isokinetic strength measurements of the hip abductor and adductor will also be assessed in a standing position.

Isometric midthigh pull (IMTP) strength test The IMTP is an isometric assessment used to determine maximal force in various athletic populations11. We will use a custom-built IMTP device that measures strength via load cells, following the principles described by Augustsson et al.10.

Lateral agility and muscular endurance Lateral agility, muscular endurance and any lower between-limb differences will be evaluated with the 30-sec Side hop test for each leg, as described5.

VO2max Peak VO2 will be performed with a graded treadmill (Rodby RL2000 60) protocol and with the player equipped with a heart rate monitor (Polar RS400; Polar, Kempele, Finland) and face mask (mask 7450 V2). Cardiorespiratory variables will be measured continuously breath-by-breath using ergospirometry (Vyntus CPX, CareFusion, Hochberg, Germany).

Speed Linear sprinting speed is assessed by three a 20-m sprint attempts using two timing gates (Witty, Microgate, Italy) with 2 minutes of recovery between each sprint.

Change of direction speed The 505 agility test will be used to assesses 180-degree turning ability using e timing gate (Witty, Microgate, Italy) as described12.

Zig-zag (running and dribbling) test The Zig-zag (running) test will be used to assess running speed with a constant change of direction using two-timing gates (Witty, Microgate, Italy) as described13.

Reactive Agility To assess football-specific agility, the reactive agility (RAG) test is used using an infrared (IR) sensor that is positioned 1.5 m from the line and a hardware module (ATMEL Corp, San Jose, CA, United States) that activates one of the four LEDs inside the 30-cm-high cones (labeled A, B, C, and D) as described14.

Neuromuscular knee control Neuromuscular knee control will be assessed and scored with one functional performance tests, the drop jump test (DJ) as described15 and video-recorded using the Coach Eye app for smart phone. To facilitate analysis and to be able to measure knee valgus coach tape will be used to mark landmarks on the SIAS, mid-patella, and mid-centered between the lateral and medial malleolus. Analysis and calculation of the valgus angle will be performed using the software program Kinovea (version 0.9.5), which is a well-established software program designed to investigate and analyze kinematic parameters.

ELIGIBILITY:
Inclusion Criteria:

* female and male academy football players aged 15-19 years and
* female and male professional football players that plays the one of the two top division in Sweden.

Exclusion Criteria:

* injuries at baseline assessment, that may affect test results

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Swedish male and female players that are playing at professional level or at academy level (from Swedish sport high schools).
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2032-01-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic endurance | Three times a year during 5 years - Change from Baseline
  VO2max performed on a treadmill measured in milliliters of oxygen per kilogram of body weight per minute (mL/kg/min).
Muscle strength | Three times a year during 5 years - Change from Baseline
  Isokinetic and isometric muscle strength of the lower extremity (m quadriceps, hamstrings, hip adduction and abduction) measured in Newton.
Sport specific performance | Three times a year during 5 years - Change from Baseline
  Speed, change of direction and agility measured in time (seconds).
Neuromuscular control | Three times a year during 5 years - Change from Baseline
  Neuromuscular control of the knee (valgus, normal, varus), measured in degrees.
Lateral agility and muscular endurance | Three times a year during 5 years - Change from Baseline
  Lateral agility, muscular endurance and any lower between-limb differences will be evaluated with the 30-sec Side hop test for each leg. Number of repetitions are measured.

SECONDARY OUTCOMES:
External training load - games and practice | Each session are reported on weekly basis during 5 years
  External training load includes; hours of training and games (unit h).
Internal training load - sRPE | Each session are reported on weekly basis during 5 years
  Estimation of session ratings of perceived exertion (sRPE) (numeric rating scale (NRS) from 0-10) after each football session.
Number of injuries | Weekly report during 5 years
  All players will report all time-loss injuries occurring during sport activity diagnosed by a physical examination, MRI, or arthroscopy. Details on injury situation, and diagnosis will be reported by the team's RPT.
Internal training load - Freshness | Weekly report during 5 years
  Freshness score will be used which includes perceived muscle soreness, sleep quality and mental stress. Each item are scored on a numeric rating scale ranging from 0-10 and a total score are calculated (0-30).

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Ryman Augustsson, PhD, Principal Investigator — Linnaeus University
Locations (1):
- Sofia Ryman Augustsson, Kalmar, Sweden

IPD SHARING:
Plan to Share IPD: No
The data will contain highly personal data from professional football players which could be traced to a specific person. These players are very sensitive because of their market value. Although de-identified, a compilation of the outcomes can reveal the person. Thus, these ethical dilemma together with the regulation on the protection of natural persons by the General Data Protection Regulation (GDPR) (2018:218), we opt not to share IPD.

REFERENCES:
- [Background] Bujnovky D, Maly T, Ford KR, Sugimoto D, Kunzmann E, Hank M, Zahalka F. Physical Fitness Characteristics of High-level Youth Football Players: Influence of Playing Position. Sports (Basel). 2019 Feb 16;7(2):46. doi: 10.3390/sports7020046. PMID 30781535
- [Background] Akbar S, Soh KG, Jazaily Mohd Nasiruddin N, Bashir M, Cao S, Soh KL. Effects of neuromuscular training on athletes physical fitness in sports: A systematic review. Front Physiol. 2022 Sep 23;13:939042. doi: 10.3389/fphys.2022.939042. eCollection 2022. PMID 36213248
- [Background] Wisloff U, Castagna C, Helgerud J, Jones R, Hoff J. Strong correlation of maximal squat strength with sprint performance and vertical jump height in elite soccer players. Br J Sports Med. 2004 Jun;38(3):285-8. doi: 10.1136/bjsm.2002.002071. PMID 15155427
- [Background] Zemkova E, Zapletalova L. The Role of Neuromuscular Control of Postural and Core Stability in Functional Movement and Athlete Performance. Front Physiol. 2022 Feb 24;13:796097. doi: 10.3389/fphys.2022.796097. eCollection 2022. PMID 35283763
- [Background] Ryman Augustsson S, Arvidsson J, Haglund E. Jump height as performance indicator for the selection of youth football players to national teams. J Sports Med Phys Fitness. 2019 Oct;59(10):1669-1675. doi: 10.23736/S0022-4707.19.09739-1. Epub 2019 May 2. PMID 31062951
- [Background] Collings TJ, Diamond LE, Barrett RS, Timmins RG, Hickey JT, DU Moulin WS, Williams MD, Beerworth KA, Bourne MN. Strength and Biomechanical Risk Factors for Noncontact ACL Injury in Elite Female Footballers: A Prospective Study. Med Sci Sports Exerc. 2022 Aug 1;54(8):1242-1251. doi: 10.1249/MSS.0000000000002908. Epub 2022 Mar 12. PMID 35320148
- [Background] Khayambashi K, Ghoddosi N, Straub RK, Powers CM. Hip Muscle Strength Predicts Noncontact Anterior Cruciate Ligament Injury in Male and Female Athletes: A Prospective Study. Am J Sports Med. 2016 Feb;44(2):355-61. doi: 10.1177/0363546515616237. Epub 2015 Dec 8. PMID 26646514
- [Background] Ryman Augustsson S, Ageberg E. Weaker lower extremity muscle strength predicts traumatic knee injury in youth female but not male athletes. BMJ Open Sport Exerc Med. 2017 Apr 16;3(1):e000222. doi: 10.1136/bmjsem-2017-000222. eCollection 2017. PMID 29259807
- [Background] Ryman Augustsson S, Gustafsson T, Ageberg E. Can tests of physical fitness predict traumatic knee injury in youth female athletes? A prospective cohort study. Phys Ther Sport. 2024 Sep;69:15-21. doi: 10.1016/j.ptsp.2024.06.007. Epub 2024 Jul 2. PMID 38991623
- [Background] Malone S, Owen A, Newton M, Mendes B, Collins KD, Gabbett TJ. The acute:chonic workload ratio in relation to injury risk in professional soccer. J Sci Med Sport. 2017 Jun;20(6):561-565. doi: 10.1016/j.jsams.2016.10.014. Epub 2016 Nov 9. PMID 27856198
- [Background] Beck NA, Lawrence JTR, Nordin JD, DeFor TA, Tompkins M. ACL Tears in School-Aged Children and Adolescents Over 20 Years. Pediatrics. 2017 Mar;139(3):e20161877. doi: 10.1542/peds.2016-1877. PMID 28228501
- [Background] Ekenros L, Friden C, von Rosen P. Does injury risk increase when youth athletes start to study at a sports high school? BMJ Open Sport Exerc Med. 2023 Nov 3;9(4):e001686. doi: 10.1136/bmjsem-2023-001686. eCollection 2023. PMID 37937308
- [Background] Fuller CW, Ekstrand J, Junge A, Andersen TE, Bahr R, Dvorak J, Hagglund M, McCrory P, Meeuwisse WH. Consensus statement on injury definitions and data collection procedures in studies of football (soccer) injuries. Br J Sports Med. 2006 Mar;40(3):193-201. doi: 10.1136/bjsm.2005.025270. PMID 16505073
- [Background] McLester CN, Nickerson BS, Kliszczewicz BM, McLester JR. Reliability and Agreement of Various InBody Body Composition Analyzers as Compared to Dual-Energy X-Ray Absorptiometry in Healthy Men and Women. J Clin Densitom. 2020 Jul-Sep;23(3):443-450. doi: 10.1016/j.jocd.2018.10.008. Epub 2018 Nov 3. PMID 30472111
- [Background] Gustavsson A, Neeter C, Thomee P, Silbernagel KG, Augustsson J, Thomee R, Karlsson J. A test battery for evaluating hop performance in patients with an ACL injury and patients who have undergone ACL reconstruction. Knee Surg Sports Traumatol Arthrosc. 2006 Aug;14(8):778-88. doi: 10.1007/s00167-006-0045-6. Epub 2006 Mar 9. PMID 16525796
- [Background] Augustsson J, Alt T, Andersson H. Speed Matters in Nordic Hamstring Exercise: Higher Peak Knee Flexor Force during Fast Stretch-Shortening Variant Compared to Standard Slow Eccentric Execution in Elite Athletes. Sports (Basel). 2023 Jul 7;11(7):130. doi: 10.3390/sports11070130. PMID 37505617
- [Background] Augustsson J, Andersson H. Differences in Peak Knee Flexor Force between Eccentric-Only and Combined Eccentric-Concentric Nordic Hamstring Exercise. Sports (Basel). 2023 Feb 7;11(2):41. doi: 10.3390/sports11020041. PMID 36828326
- [Background] Falk Neto JH, Tibana RA, de Sousa NMF, Prestes J, Voltarelli FA, Kennedy MD. Session Rating of Perceived Exertion Is a Superior Method to Monitor Internal Training Loads of Functional Fitness Training Sessions Performed at Different Intensities When Compared to Training Impulse. Front Physiol. 2020 Aug 12;11:919. doi: 10.3389/fphys.2020.00919. eCollection 2020. PMID 32903483
- [Background] Waiteman MC, Garcia MC, Briani RV, Norte G, Glaviano NR, De Azevedo FM, Bazett-Jones DM. Can Clinicians Trust Objective Measures of Hip Muscle Strength From Portable Dynamometers? A Systematic Review With Meta-analysis and Evidence Gap Map of 107 Studies of Reliability and Criterion Validity Using the COSMIN Methodology. J Orthop Sports Phys Ther. 2023 Nov;53(11):655-672. doi: 10.2519/jospt.2023.12045. PMID 37787581
- [Background] Augustsson J, Gunhamn T, Andersson H. An Assessment of the Ratio between Upper Body Push and Pull Strength in Female and Male Elite Swedish Track and Field Throwers. Sports (Basel). 2024 Jul 24;12(8):201. doi: 10.3390/sports12080201. PMID 39195577
- [Background] Giles G, Lutton G, Martin J. Scoping Review of the Isometric Mid-Thigh Pull Performance Relationship to Dynamic Sport Performance Assessments. J Funct Morphol Kinesiol. 2022 Dec 15;7(4):114. doi: 10.3390/jfmk7040114. PMID 36547660
- [Background] Faltstrom A, Hagglund M, Hedevik H, Lindblom H, Kvist J. The side hop test: Validity, reliability, and quality aspects in relation to sex, age and anterior cruciate ligament reconstruction, in soccer players. Phys Ther Sport. 2023 Jul;62:39-45. doi: 10.1016/j.ptsp.2023.05.008. Epub 2023 Jun 3. PMID 37300972
- [Background] Altmann S, Ringhof S, Neumann R, Woll A, Rumpf MC. Validity and reliability of speed tests used in soccer: A systematic review. PLoS One. 2019 Aug 14;14(8):e0220982. doi: 10.1371/journal.pone.0220982. eCollection 2019. PMID 31412057
- [Background] Emmonds S, Nicholson G, Begg C, Jones B, Bissas A. Importance of Physical Qualities for Speed and Change of Direction Ability in Elite Female Soccer Players. J Strength Cond Res. 2019 Jun;33(6):1669-1677. doi: 10.1519/JSC.0000000000002114. PMID 28723816
- [Background] Wragg CB, Maxwell NS, Doust JH. Evaluation of the reliability and validity of a soccer-specific field test of repeated sprint ability. Eur J Appl Physiol. 2000 Sep;83(1):77-83. doi: 10.1007/s004210000246. PMID 11072777
- [Background] Pojskic H, Aslin E, Krolo A, Jukic I, Uljevic O, Spasic M, Sekulic D. Importance of Reactive Agility and Change of Direction Speed in Differentiating Performance Levels in Junior Soccer Players: Reliability and Validity of Newly Developed Soccer-Specific Tests. Front Physiol. 2018 May 15;9:506. doi: 10.3389/fphys.2018.00506. eCollection 2018. PMID 29867552
- [Background] Augustsson SR, Nae J, Karlsson M, Peterson T, Wollmer P, Ageberg E. Postural orientation, what to expect in youth athletes? A cohort study on data from the Malmo Youth Sport Study. BMC Sports Sci Med Rehabil. 2021 Jul 24;13(1):76. doi: 10.1186/s13102-021-00307-y. PMID 34301323
- See also: Related Info — https://lnu.se/en/research/research-projects/project-sustainable-football/

DOCUMENTS (2):
  • Statistical Analysis Plan (2024-07-28): https://cdn.clinicaltrials.gov/large-docs/84/NCT07325084/SAP_000.pdf
  • Informed Consent Form (2024-08-31): https://cdn.clinicaltrials.gov/large-docs/84/NCT07325084/ICF_001.pdf